CLINICAL TRIAL: NCT05769010
Title: A Prospective, Open-label Explorative Study of SHR-A1811 in HER2-expression Advanced Breast Cancer with Brain Metastases
Brief Title: Study of SHR-A1811 in HER2-expression Advanced Breast Cancer with Brain Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Min Yan, MD, Chief Physician, Henan Cancer Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HNCH-MBC12; HNCH-MBC12-BM04 (Other: Henan Cancer Hospital)
Record Dates: First submitted 2023-03-02; First posted 2023-03-15 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Arm 1 (Experimental): HER2-positive: SHR-A1811
  Interventions: Drug: SHR-A1811
- Arm 2 (Experimental): HER2-positive: SHR-A1811 and pyrotinib
  Interventions: Drug: SHR-A1811; Drug: Pyrotinib
- Arm 3 (Experimental): HER2-positive: SHR-A1811 and bevacizumab
  Interventions: Drug: SHR-A1811; Drug: Bevacizumab
- Arm 4 (Experimental): HER2-low: SHR-A1811
  Interventions: Drug: SHR-A1811
- Arm 5 (Experimental): HER2-low: SHR-A1811 and bevacizumab
  Interventions: Drug: SHR-A1811; Drug: Bevacizumab

INTERVENTIONS:
Drug: SHR-A1811 — SHR-A1811: intravenous
Drug: Pyrotinib — Pyrotinib: oral
  Arms: Arm 2
Drug: Bevacizumab — Bevacizumab: intravenous
  Arms: Arm 3; Arm 5

SUMMARY:
This study aimed to evaluate the use of SHR-A1811 in HER2-expression Advanced Breast Cancer patients with brain metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Females ≥18 yrs old;
2. Pathologically confirmed HER2-positive or HER2-low advanced breast cancer;
3. At least one measurable intracranial lesion according to RANO-BM criteria, which had not received local treatment;
4. Without prior cranial radiation and had no indication for immediate local treatment or refuse to local treatment;
5. More than 2 weeks from last systemic treatment; patients with new brain lesions after craniocerebral surgery were admitted if no radiotherapy was performed. Patients with HER2-Low disease must not have systemic treatment for brain metastases.
6. Prior HER2-target treatment, endocrine therapy and chemotherapy was allowed;
7. Life expectancy is not less than 6 months.
8. Adequate function of major organs.

Exclusion Criteria:

1. Leptomeningeal involvement;
2. CNS complications requiring emergency neurosurgical intervention (e.g. excision, shunt tube placement);or uncontrolled symptomatic brain metastases;
3. Previous treatment with trastuzumab deruxtecan (DS-8201a) or any other antibody drug conjugate (ADC) which consists of an exatecan derivative that is a topoisomerase 1 inhibitor;
4. Patients who had progressed on previous HER2 tyrosine kinase inhibitor therapy were excluded from Arm 2, and those who had progressed on previous bevacizumab therapy were excluded from Arm 3;
5. No concurrent antitumor therapy for metastatic cancer other than the study treatment;
6. Antitumor radiotherapy, chemotherapy, surgery, targeted therapy, or immunotherapy within 2 weeks or endocrine therapy within 1 week prior to enrolment;
7. Participated in other drug clinical trials within 4 weeks before admission;
8. History of clinically significant lung disease；
9. Other malignant tumors, excluding cured cervical carcinoma in situ, skin basal cell carcinoma or skin squamous cell carcinoma, have been diagnosed in the past five years.
10. According to the judgement of the researchers, there are concomitant diseases that seriously endanger the safety of patients or affect the completion of research (including, but not limited to, severe hypertension, severe diabetes, active infections, etc.).
11. Any other conditions that researchers believe that patients are unsuitable for this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
CNS-ORR by investigator | 2 months
  CNS-ORR was defined as percentage of participants with CNS response assessed by the investigator according to RANO-BM criteria

SECONDARY OUTCOMES:
ORR by investigator using RECIST Guideline (Version 1.1) | 2 months
  ORR was defined as percentage of participants with best (confirmed) overall response (BOR) of either CR or PR assessed by the investigator according to RECIST version 1.1
PFS | up to 1.5 years
  PFS was defined as the time from first dose to first documented disease progression (PD) or death from any cause, whichever occurred first
Adverse events | up to 1.5 years
  Proportion of participants experienced adverse events during the study period

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No